CLINICAL TRIAL: NCT06079632
Title: Telehealth Parent Coaching to Improve Activity Participation for Young Children With Autism Spectrum Disorder and Sensory Processing Disorders: A Prospective Study
Brief Title: Telehealth Parent Coaching to Improve Activity Participation for Young Children With ASD and SPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency); National Taiwan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202301189RINA
Record Dates: First submitted 2023-09-28; First posted 2023-10-12 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Sensory Processing Disorder; Autism Spectrum Disorder
Keywords: Sensory Processing Disorder; Parent-mediated intervention; Autism Spectrum Disorder; Parent Coaching via Telehealth
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: In the first experiment, multiple baseline design will be used to examine the feasibility of the interventions. Each participant will first receive parent-child interaction strategy coaching every week via Telehealth, followed by sensory processing strategy coaching (C1) provided every week via Telehealth. In the second experiment, RCT design will be applied to explore the efficacy of the interventions. Participants will be randomly allocated to the treatment group or the control group. The intervention group will receive weekly, one-on-one parent-child interaction and sensory processing strategy coaching via Telehealth for 12 weeks. The control group will be provided with weekly self-learning materials and group discussion session for 12 weeks. Measures will be taken at pre-test, post-test, and 3-month follow-up.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single subject experiment (Experimental): Each participant will first receive one-hour, one-on-one parent-child interaction strategy coaching every week via Telehealth until the parent's parent-child interaction skills and the child's social communication abilities reach a stable or upward trend, and the parent's sensory processing strategy utilization ability and the child's daily life participation scores that are continuously collected shows a stable or downward trend. After which, the one-hour, one-on-one sensory processing strategy coaching (C1) will be provided every week via Telehealth until the parent's sensory processing strategy utilization ability and the child's activity participation level reaches a stable trend.
  Interventions: Behavioral: parent coaching via telehealth
- RCT, Treatment group (Experimental): Participant receive 12 weeks of sensory processing strategy coaching and parent-child interaction strategy coaching intervention.
  Interventions: Behavioral: parent coaching via telehealth
- RCT, Active Comparator (Active Comparator): Participant will be provided with weekly self-learning materials and group discussion session for 12 weeks.
  Interventions: Behavioral: weekly self-learning materials and group discussion session

INTERVENTIONS:
Behavioral: parent coaching via telehealth — Participants receive 12 weeks of parent-child interaction strategy coaching and sensory processing strategy coaching intervention.
  Arms: RCT, Treatment group; Single subject experiment
Behavioral: weekly self-learning materials and group discussion session — Participants receive 1-hour self-learning materials, including parent-child interaction and sensory processing strategies, and 1-hour remote group discussion session weekly.
  Arms: RCT, Active Comparator

SUMMARY:
This clinical trial aims to develop parent-child interaction strategy coaching and sensory processing strategy coaching via Telehealth and examine the feasibility and efficacy of the interventions in young children with autism spectrum disorder who have sensory processing disorder.

In the first experiment, the investigators will apply a single-subject research design and one-group pre-post test design to explore the feasibility of the coaching interventions. In the second experiment, RCT design will be used to examine the effectiveness of parent coaching. Sixty-five children with ASD and their parents will be randomly assigned to the intervention or control group. The intervention group will receive weekly parent-child interaction and sensory processing strategy coaching for 12 weeks. The control group will be provided with weekly self-learning materials and group discussion session for 12 weeks. Additionally, the follow-up test will be administered three months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* The child is 3 to 5 years old
* The child is diagnosed with ASD by a child psychiatrist or specialist in psychology based on the DSM-5's diagnostic criteria
* The child's score falls within the category of dysfunction in one or more sensory processing functions in the Sensory Profile (3-10 years old version)

Exclusion Criteria:

* Children diagnosed with major neuromuscular dysfunction or other disease diagnoses, such as epilepsy or other genetic diseases
* Children whose parents could not speak Hokkenese or Chinese and read in Chinese
* Individuals who have participated in the first year of this study

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The performance and satisfaction with the child's daily participation | up to 25 weeks
  Measured by the Canadian Occupational Performance Measure in the RCT experiment. The score could range from 1 to 10, with higher scores implied greater performance and higher satisfaction with the child's daily participation.
The parent's parent-child interaction strategy utilization | through study completion, an average of 4 months
  Measured by the self-developed measurement - the Parental Parent-Child Interaction Strategy Rating Scale in the single subject experiment. The score could range from 20 to 80, with higher scores implied greater parent-child interaction strategy utilization.
The child's social communication ability | through study completion, an average of 4 months
  Measured by the self-developed measurement - the Social Communication Rating Scale for young children in the single subject experiment. The score could range from 0 to 38, with higher scores implied greater social communication ability.

SECONDARY OUTCOMES:
The social functioning and adaptive behavior of the child | up to 25 weeks
  Measured by the Vineland Adaptive Behavior Scales - Third Edition in the RCT experiment. The score could range from 20 to 160, with higher scores implied greater social functioning and adaptive behavior.
The attainment of the selected goal related to issues with the child's sensory processing disorder | up to 25 weeks
  Measured by the Goal Attainment Scale in the RCT experiment. The score could range from -2 to 2, with higher scores implied greater attainment of the selected goal related to issues with the child's sensory processing disorder.
The attainment of the selected goal related to issues with the child's sensory processing disorder | through study completion, an average of 4 months
  Measured by the Goal Attainment Scale in the single subject experiment. The score could range from -2 to 2, with higher scores implied greater attainment of the selected goal related to issues with the child's sensory processing disorder.
The child's performance in social communication | up to 25 weeks
  Measured by the Brief Observation of Social Communication Change in the RCT experiment. The score could range from 0 to 85, with higher scores implied greater social communication performance.
The parent's self-perceived parental competence | up to 25 weeks
  Measured by the Parenting Sense of Competence Scale in the RCT experiment. The score could range from 17 to 102, with higher scores implied greater self-perceived parental competence.
The parent's self-perceived parental competence | through study completion, an average of 4 months
  Measured by the Parenting Sense of Competence Scale in the single subject experiment. The score could range from 17 to 102, with higher scores implied greater self-perceived parental competence.
The parent's self-perceived stress within the family system | up to 25 weeks
  Measured by the Parenting Stress Index - Short Form in the RCT experiment. The score could range from 35 to 175, with higher scores implied greater self-perceived stress within the family system
The parent's self-perceived life quality within the last two weeks | up to 25 weeks
  Measured by the WHOQOL-BREF - Taiwan version in the RCT experiment. The score could range from 4 to 20 in each domain, with higher scores implied greater self-perceived life quality within the last two weeks
The child's social communication ability | up to 25 weeks
  Measured by the self-developed measurement - the Social Communication Rating Scale for young children in the RCT experiment. The score could range from 0 to 38, with higher scores implied greater social communication ability
The parent's parent-child interaction strategy utilization | up to 25 weeks
  Measured by the self-developed measurement - the Parental Parent-Child Interaction Strategy Rating Scale in the RCT experiment. The score could range from 20 to 80, with higher scores implied greater parent-child interaction strategy utilization.
The performance and satisfaction with the child's daily participation | through study completion, an average of 4 months
  Measured by the Canadian Occupational Performance Measure in the single subject experiment. The score could range from 1 to 10, with higher scores implied greater performance or higher satisfaction with the child's daily participation.

OTHER OUTCOMES:
The parent's satisfaction with the online intervention | 1 week
  Measured by self-developed questionnaire used to assess parental parent's satisfaction with the online intervention in the RCT experiment. The score could range from 17 to 68, with higher scores implied higher satisfaction with the online intervention.
The parent's satisfaction with the online intervention | 1 week
  Measured by self-developed questionnaire used to assess parental parent's satisfaction with the online intervention in the single subject experiment. The score could range from 17 to 68, with higher scores implied higher satisfaction with the online intervention.
The coach's satisfaction with the online intervention | 1 week
  Measured by self-developed questionnaire used to assess the coach's satisfaction with the online intervention in the RCT experiment. The score could range from 11 to 44, with higher scores implied higher satisfaction with the online intervention.
The coach's satisfaction with the online intervention | 1 week
  Measured by self-developed questionnaire used to assess the coach's satisfaction with the online intervention in the single subject experiment. The score could range from 11 to 44, with higher scores implied higher satisfaction with the online intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Hui Tseng, phD, Principal Investigator — National Taiwan University